CLINICAL TRIAL: NCT00551434
Title: Effect of Creatine and L-Arginine on Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Effect of Creatine and L-Arginine on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-22852
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Creatine; Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Dietary Supplement: Creatine
- 2 (Experimental)
  Interventions: Dietary Supplement: l-arginine
- 3 (Experimental)
  Interventions: Dietary Supplement: L-arginine and creatine
- 4 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo, double

INTERVENTIONS:
Dietary Supplement: Creatine — Creatine 21 g daily
  Arms: 1
Dietary Supplement: L-arginine and creatine — L-arginine
  Arms: 3
Dietary Supplement: l-arginine — l-arginine 9 g daily
  Arms: 2
Dietary Supplement: placebo, double — placebo
  Arms: 4

SUMMARY:
The study is a double blind 2x2 factorial study. Patients with coronary disease will be randomly be assigned to L-arginine (9 g/day), creatine 21 g/d, both, or neither dietary supplement. The function of the endothelium will be tested using ultrasound before and after each treatment. These studies will help us understand why the endothelium is abnormal in patients with coronary artery disease and how L-arginine is acting on endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease

Exclusion Criteria:

* Pregnancy
* Creatine use within one month of study
* L-arginine use within one month of study
* Change in dose or initiation of lipid lowering therapy, aspirin therapy, or angiotensin converting enzyme therapy within one month of study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2002-08; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 5 days

SECONDARY OUTCOMES:
serum arginine, creatine, creatinine, homocysteine | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston Medical Center